CLINICAL TRIAL: NCT04157985
Title: Evaluating Length of Treatment With PD-1/PD-L1 Inhibitor in Advanced Solid Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dan Zandberg (Other)
Responsible Party: Sponsor-Investigator, Dan Zandberg, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 19-135
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors; NSCLC; Bladder Cancer; HNSCC; Renal Cancer; Melanoma; Anal Cancer; Colorectal Cancer; Cholangiocarcinoma; Gastric Cancer; Hepatocellular Carcinoma; Merkel Cell Carcinoma; Cervical Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Squamous Cell Carcinoma of Head and Neck; Kidney Neoplasms; Melanoma; Anus Neoplasms; Colorectal Neoplasms; Cholangiocarcinoma; Stomach Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Merkel Cell; Uterine Cervical Neoplasms | interventions — pembrolizumab; Nivolumab; atezolizumab; Ipilimumab; cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continue Treatment with PD-1/PD-L1 inhibitor (Active Comparator): Continued standard of care treatment with PD-1/PD-L1 -1 checkpoint inhibitor after 12 months of checkpoint inhibitor treatment.
  Interventions: Drug: Continue PD-1/PD-L1 Inhibitors treatment
- Discontinue Treatment with PD-1/PD-L1-1 inhibitor (Experimental): Discontinued standard of care treatment with PD-1/PD-L1 -1 checkpoint inhibitor after 12 months of checkpoint inhibitor treatment.
  Interventions: Other: Discontinue PD-1/PD-L1-1 inhibitor

INTERVENTIONS:
Drug: Continue PD-1/PD-L1 Inhibitors treatment — Continued treatment with PD-1/PD-L1-1 inhibitor
  Other Names: Keytruda (pembrolizumab); Optiva (nivolumab); Tecentriq (atezolizumab); Yervoy (ipilimumab); LIBTAYO (cemiplimab)
  Arms: Continue Treatment with PD-1/PD-L1 inhibitor
Other: Discontinue PD-1/PD-L1-1 inhibitor — Discontinued treatment with PD-1/PD-L1-1 inhibitor
  Arms: Discontinue Treatment with PD-1/PD-L1-1 inhibitor

SUMMARY:
Based on the overwhelming positive response to this survey and the large number of patients being treated with PD-1/PD-L1 therapy in the UPMC system, the investigators are proposing a trial that will randomize patients who have disease stability to stop treatment at 1 year or continue treatment until disease progression. The investigators anticipate that the results of this study will answer questions regarding the optimal duration of treatment. therapy.

DETAILED DESCRIPTION:
Within the UPMC system, approximately 2,300 patients received PD-1/PD-L1 therapy for a variety of advanced solid tumors within the past year. It is anticipated that this number will increase as the clinical indications for treatment with these agents also increase. The investigators conducted a survey of 60 Medical Oncologists within the UPMC system regarding their interest in a trial that will attempt to address the question of optimal length of PD-1/PD-L1 treatment. Fifty-two (86.7%) physicians indicated that they would participate in a clinical trial that had a primary goal of determining whether it was feasible to stop immunotherapy after 1 year of treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have an advanced solid tumor malignancy (specifically NSCLC, bladder, HNSCC, renal, melanoma, cervical, Merkel cell, MMR/MSI [colon, rectal, cholangio, esophageal, ovarian, uterine], anal, gastric and GE junction, hepatocellular, triple negative breast cancer) that is being treated with a PD-1/PD-L1 inhibitor including pembrolizumab, nivolumab, atezolizumab, durvalumab, or avelumab according to standard of care treatment.
* Patients who initially started treatment with another agent in combination with the PD-1/PD-L1 inhibitor, i.e. chemotherapy, ipilumumab, are eligible.
* Patients must have at least stable disease as evidenced by scans performed within 6 weeks of randomization.
* Signed Informed consent allowing randomization to stopping immunotherapy at 1 year ± 6 weeks versus continued treatment beyond 1 year.
* Patients can have measurable or non-measurable disease per RECIST v1.1.
* Patients cannot be enrolled in a clinical trial.

Exclusion Criteria:

* Patients with documented progressive disease prior to randomization.
* Patients with an immune-related toxicity preventing the continuation of treatment beyond 1 year at the treating physician's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Time to next treatment | Up to 36 months
  In patients who have already been treated with a PD-1 or PD-L1 inhibitor for one year, the difference in progression-free survival (time to next treatment, progression or death, whichever occurs first) between patients who stop treatment and patients who continue treatment.
Progression-free Survival (PFS) (at between 2-3.9 months) | Between 2 months and 3.9 months
  The (median) length of time from the initial date of treatment to the date of documented progression, or the date of death due to any cause (in the absence of progression, whichever occurs first), with progression defined by RECIST v1.1.Per RECIST v1.1, progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least5mm. For non-target lesions, PD: Unequivocal progression of existing non-target lesions. The appearance of one or more new lesions is also considered progression.
Progression-free Survival (PFS) (at between 4-7.9 months) | Between 4 months and 7.9 months
  The (median) length of time from the initial date of treatment to the date of documented progression, or the date of death due to any cause (in the absence of progression, whichever occurs first), with progression defined by RECIST v1.1.Per RECIST v1.1, progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least5mm. For non-target lesions, PD: Unequivocal progression of existing non-target lesions. The appearance of one or more new lesions is also considered progression.
Progression-free Survival (PFS) | Up to 36 months
  The (median) length of time from the initial date of treatment to the date of documented progression, or the date of death due to any cause (in the absence of progression, whichever occurs first), with progression defined by RECIST v1.1.Per RECIST v1.1, progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least5mm. For non-target lesions, PD: Unequivocal progression of existing non-target lesions. The appearance of one or more new lesions is also considered progression.

SECONDARY OUTCOMES:
Incidence of irAEs (Immune-Related Adverse Events) | Up to 36 months
  Proportion of participants in a disease stratum and treatment arm who experience at least one AE of any grade (per Common Terminology Criteria for Adverse Events (CTCAE v5.0)), at least possibly related to treatment in the categories of colitis, hepatitis, pnemonitis, hypophysitis or hypopituitarism, hypothyroidism, fatigue, diarrhea, rash, arthritis, arthralgia, back pain, musculoskeletal pain or myalgia, or any other category that is felt to be related to treatment.
Overall Survival (OS) | Up to 36 months
  The length of time from the start of treatment that patients are still alive.
Best Objective Response (BOR) | Up to 36 months
  Proportions of participants who restart for disease progression in each disease stratum, who experience a best objective response (progressive disease, stable disease, partial response, complete response) per RECIST v1.1 (Response Evaluation Criteria in Solid Tumors);Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (target or non-target) with reduction in short axis to <10 mm;Partial Response (PR): ≥ 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters;Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, (reference smallest sum diameters);Progressive Disease (PD): ≥ 20% increase in the sum of diameters of target lesions (reference smallest sum diameters); the sum must also demonstrate an absolute increase of at least 5 mm; (appearance ≥ 1 new lesions is considered progression).

CONTACTS AND LOCATIONS:
Overall Officials: Dan Zandberg, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No